CLINICAL TRIAL: NCT06888934
Title: Evaluation of the Treatment of Arthritis and the Correction of Bone Alignment Default of the Toes Using the Lync® Medical Device
Brief Title: Evaluation of the Treatment of Arthritis and the Correction of Bone Alignment Default of the Toes With Lync
Acronym: LYNC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Novastep (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024-1
Record Dates: First submitted 2025-03-04; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Arthritis Foot; Bone Alignment Defaults
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention with Lync device (Experimental): One arm in the study : treatment of arthritis and/or correction of bone alignement default in the toes (mallet toes, claw toes, hammer toes) wwith Lync device.
  Interventions: Device: Intervention with Lync device.

INTERVENTIONS:
Device: Intervention with Lync device. — Treatment of arthritis and/or correction of bone alignement default in the toes (mallet toes, claw toes, hammer toes) with Lync device.

SUMMARY:
The "LYNC" clinical investigation aims to confirm the clinical benefits, performance and safety of the Lync® device when implanted in the toes for the treatment of arthritis and correction of bone misalignments.

The main objective of the study is to confirm the clinical benefits of the Lync® device for the treatment of arthritis and the correction of bone alignment default, by evaluating the restoration of the functional capacities of the forefoot at 3 -4 months post-operative follow-up with AOFAS-LMIS score.

DETAILED DESCRIPTION:
The clinical evaluation demonstrates that the clinical benefits, performance and safety of the Lync® device when implanted in the toes for the treatment of arthritis are not covered by any clinical data on similar devices.

The "LYNC" clinical investigation aims to confirm the clinical benefits, performance and safety of the Lync® device on 76 cases (feet) when implanted in the toes for the treatment of arthritis and correction of bone misalignments.

The main objective of the study is to confirm the clinical benefits of the Lync® device for the treatment of arthritis and the correction of bone alignment default, by evaluating the restoration of the functional capacities of the forefoot at 3 -4 months post-operative follow-up with AOFAS-LMIS score as primary endpoint.

The secondary objectives of the study are:

* To confirm the clinical benefits of the Lync® device for the treatment of arthritis and the correction of bone alignment default in the toes, by evaluating the reduction in patient pain during the 3-4 month postoperative visit.
* To confirm the clinical performance of the Lync® device for the treatment of arthritis and the correction of bone alignment default in the toes, by evaluating the radiographic parameters (bone consolidation) during the 3-4 month postoperative visit.
* To confirm the safety of the Lync® device for the treatment of arthritis and the correction of bone alignment default in the toes, by evaluating the occurrence of adverse events, complications and device defects at the various postoperative follow-up visits.

The secondary endpoints associated with the secondary objective are:

* The change in the VAS score will be evaluated at the postoperative visit at 3-4 months compared to that at the preoperative visit.
* The assessment of bone consolidation will be carried out at the post-operative visit at 3-4 months. An additional visit at 6 months, assessing bone union, will be carried out ifbone union has not occurred 3-4 months post-operatively, in accordance with theinvestigators' current practice.
* The collection of adverse events and defects will be done throughout the follow-up by the surgeons thanks to questioning of the patient, assessments of clinical and radiographic examinations of the foot.

ELIGIBILITY:
Inclusion Criteria:

* Patient requiring treatment of arthritis and/or correction of bone alignement defaultin the toes (mallet toes, claw toes, hammer toes),
* Use of the Lync® intramedullary osteosynthesis implantable medical device,
* No associated surgical procedures except:▪Flexor release/tenotomy

  * MTP Arthrolysis / Extensor Lengthening
  * Tendon transfers
  * Phalangeal osteotomy
* Adult patient,
* Patient capable of respecting the prescriptions and recommendations of his surgeon,
* Patient able to read and understand the information note and the consent form,
* Patient able to sign a consent form.

Exclusion Criteria:

* Patient presenting a contraindication to the device under investigation;
* Simultaneous participation in another clinical investigation protocol;
* Adults subject to legal protection (judicial protection, curatorship, guardianship),persons deprived of their liberty, pregnant or breastfeeding women, minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
EFAS (EUROPEAN FOOT AND ANKLE SOCIETY) score | 3 to 4 post-operative months
  Score of functional capacities of the forefoot at 3-4 post-operative months thanks to EFAS score (EUROPEAN FOOT AND ANKLE SOCIETY score : quality of life questionnaire). This six-item scale measures pain and physical function.
  The maximum score is 24 points (best possible) and the minimum score is 0 poins (worst possible).

SECONDARY OUTCOMES:
VAS (Visual Analogue Scale) pain score | 3 to 4 post-operative months
  Reduction in patient pain with VAS pain score (Visual Analogue Scale for pain) at 3-4 post-operative months.
  The maximum score is 10 points (maximum pain) and the minimum score is 0 poins (minimal pain).
Bone consolidation | 3 to 4 post-operative months
  Radiographic parameters: bone consolidation or no bone consolidation according to the surgeon, at 3-4 post-operative months.
occurrence of adverse events, complications, device defects | through study completion, an average of 6 months
  Safety evaluated with occurrence (number and description) of adverse events, complications and device defects throughout the study (maximum 6 post-operative months)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Clinique Saint-Charles, Lyon
  - Polyclinique du Val de Saône, Mâcon
  - Centre Chirurgical ADR, Nancy
  - Clinique Mutualiste Catalane, Perpignan
  - Polyclinique Lyon Nord, Rillieux-la-Pape

IPD SHARING:
Plan to Share IPD: No